CLINICAL TRIAL: NCT04259138
Title: VERDICT: In actiVE Ulcerative Colitis, a RanDomIzed Controlled Trial for Determination of the Optimal Treatment Target
Brief Title: Determination of the Optimal Treatment Target in Ulcerative Colitis
Acronym: VERDICT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alimentiv Inc. (Other)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP1706; 2019-002485-12 (EudraCT Number)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Intervention Model Description: In this study, participants with active UC will be randomized in a 5:4:1 ratio (initially 2:3:5) to 1 of 3 treatment target groups. Participants will be assigned a treatment algorithm based on their existing UC treatment at time of entry. Treatment algorithms may include the use of vedolizumab. A key premise is that vedolizumab has a favorable safety profile and can be used to treat participants who are in symptomatic remission but who have not attained endoscopic or histopathologic remission.
  Participants will be assessed to determine it remission target is achieved at weeks 16, 32 and 48. If the participant has achieved their treatment target, they will continue that line of therapy. If the participant has not achieved their treatment target, treatment and/or dose escalation will be administered according to the algorithm.
Who Masked: Participant
Masking Description: Investigators will be trained on the treatment algorithms and target groups. Study participants will be blinded to target group assignment, whereas investigators will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Symptomatic remission (Other): Treatment target defined as achievement of corticosteroid-free symptomatic remission.
  Interventions: Biological: Treatment Algorithm A; Biological: Treatment Algorithm B; Biological: Treatment Algorithm C
- Symptomatic and endoscopic remission (Other): Treatment target defined as achievement of corticosteroid-free symptomatic remission plus endoscopic remission.
  Interventions: Biological: Treatment Algorithm A; Biological: Treatment Algorithm B; Biological: Treatment Algorithm C
- Symptomatic, endoscopic and histological remission (Other): Treatment target defined as achievement of corticosteroid-free symptomatic remission plus endoscopic remission plus histological remission.
  Interventions: Biological: Treatment Algorithm A; Biological: Treatment Algorithm B; Biological: Treatment Algorithm C

INTERVENTIONS:
Biological: Treatment Algorithm A — Participants who are not on UC treatment at screening (or who have only used topical therapy) will require standard first-line therapy. Either oral 5-ASA and/or immunosuppressive (azathioprine, 6-mercaptopurine, or methotrexate), with optional oral corticosteroid up to a maximum of 30 mg or prednisone or equivalent, will be initiated.
  Other Names: vedolizumab
Biological: Treatment Algorithm B — Participants who are taking oral 5-ASA, immunosuppressive (azathioprine, 6-mercaptopurine, methotrexate), and/or oral corticosteroid at screening will follow the treatment algorithm.
  Participants will change to intravenous vedolizumab therapy.
  Participants will be assessed to determine it remission target is achieved at weeks 16, 32 and 48. If the participant has achieved their treatment target, they will continue that line of therapy. If the participant has not achieved their treatment target, treatment and/or dose escalation will be administered according to the algorithm.
  Other Names: vedolizumab
Biological: Treatment Algorithm C — Participants who are taking a TNFα antagonist (infliximab, golimumab, or adalimumab), tofacitinib, or ustekinumab therapy at screening will follow the treatment algorithm.
  Participants will change to intravenous vedolizumab therapy.
  Participants will be assessed to determine it remission target is achieved at weeks 16, 32 and 48. If the participant has achieved their treatment target, they will continue that line of therapy. If the participant has not achieved their treatment target, treatment and/or dose escalation will be administered according to the algorithm.
  Other Names: vedolizumab

SUMMARY:
Disease activity and response to therapy in ulcerative colitis (UC) can be assessed by a range of endpoints including symptoms, endoscopic mucosal activity, histological disease activity, and biomarkers. This study aims to determine the optimal treatment target, which is a research priority for the management of UC both to inform clinical practice and to help inform regulatory endpoints and targets for drug development.

Participants with active UC will be randomized in a 5:4:1 (initially 2:3:5) ratio to 1 of 3 groups, each with a different treatment target. Treatment targets will be defined as:

* Group 1: corticosteroid-free symptomatic remission
* Group 2: corticosteroid-free endoscopic + symptomatic remission
* Group 3: corticosteroid-free histological + endoscopic + symptomatic remission

An interim analysis was performed to assess the proportion of subjects that reached their assigned treatment target after 50 subjects in each group had reached the first 32-week assessment. The interim analysis and projections made based on target achievement rates for all subjects included in the interim analysis resulted in a recommendation to adjust the randomization ratio from 2:3:5 to 5:4:1 for Groups 1, 2 and 3 respectively as of May 5th, 2023. This change was necessary in order to complete the study with approximately 100 subjects achieving treatment target within each group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosis of UC confirmed by clinical, endoscopic, and histological evidence prior to screening as per standard criteria.
3. Moderately to severely active UC with a Mayo rectal bleeding subscore ≥ 1 and a MES ≥ 2, with minimum disease extent of 15 cm and objective evidence of inflammation that can be visualized using central endoscopic imaging system.
4. Ability of participant to participate fully in all aspects of this clinical trial.
5. Written informed consent must be obtained and documented.
6. Agree not to participate in an investigational trial for the duration of the trial (observation or other noninterventional trials may be permitted at the discretion of the investigator).
7. Negative standard of care tuberculosis (TB) test and hepatitis B and C test prior to randomization unless negative results available from within 12 months prior.
8. A male participant who is nonsterilized* and sexually active with a female partner of childbearing potential* agrees to use adequate contraception* from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.
9. A female participant of childbearing potential* who is sexually active with a nonsterilized* male partner agrees to use routinely adequate contraception* from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.
10. Up to date with colorectal carcinoma surveillance according to local standards and guidelines. If a subject is not up to date at screening, a standard of care surveillance assessment may be performed during the screening period.
11. Participants who are not responding to their existing treatment for UC (Netherlands-specific criterion).

Exclusion Criteria:

1. Participants who have historically failed (i.e., had an inadequate response with, lost response to, or were intolerant to) 2 or more compounds or classes of advanced therapeutic options (biologics or small molecules; e.g., anti-TNFs, ustekinumab, or tofacitinib) for the treatment of their UC.
2. Current or previous treatment with vedolizumab, etrolizumab, or natalizumab.
3. Topical therapy (corticosteroid or 5-aminosalicylate [5-ASA]) use within 2 weeks prior to screening endoscopy.
4. Change to oral corticosteroid dosing within 2 weeks prior to randomization or a corticosteroid dose of > 30 mg of prednisone or equivalent at randomization.
5. Known diagnosis of CD, indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic colitis.
6. Short gut syndrome.
7. Positive stool culture for or active Clostridioides difficile infection (as demonstrated by positive toxin and/or antigen).
8. Known hepatitis B or C infection. If a negative test result is available in the 12 months prior to randomization, retesting is not required.
9. Known active or latent TB; if a negative test result is available in the 12 months prior to randomization, confirmatory testing (per standard of care) is not required before randomization.
10. Received any investigational drug within 30 days prior to randomization/target assignment.
11. Serious underlying disease other than UC that in the opinion of the investigator may interfere with the participant's ability to participate fully in the study or would compromise participant safety (such as history of malignancies, major neurological disorders, or any unstable or uncontrolled medical disorder).
12. History of alcohol or drug abuse that in the opinion of the investigator may interfere with the participant's ability to comply with the study procedures.
13. The participant has active cerebral/meningeal disease, signs, symptoms, or any history of progressive multifocal leukoencephalopathy (PML) prior to randomization.
14. Hypersensitivity to any excipient of vedolizumab.
15. Active severe infection such as sepsis, cytomegalovirus, listeriosis, or opportunistic infection.
16. History of HIV or positive test at screening (Italy-specific criterion).
17. Any other contraindication(s)to vedolizumab (Italy-specific criterion).
18. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 18 weeks after the last dose; or intending to donate ova during such time period.
19. If male, the participant intends to donate sperm during the course of this study or for 18 weeks after the last dose.
20. Vaccination with a live or live-attenuated vaccine within 4 weeks prior to randomization, or planned vaccination during conduct of the study, except vaccination for coronavirus disease of 2019 (COVID-19).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Time to UC-related Complication Between Treatment Target Groups 1 and 3 | From date of treatment target achievement until date of first UC-related complication until end of study (Week 96), whichever came first
  Time to UC-related complication starting when a participant reaches their assigned treatment target, compared between treatment target groups 1 and 3.

SECONDARY OUTCOMES:
Difference in Time to UC-related Complication Compared Between Treatment Target Groups 1 and 2. | From date of treatment target achievement until date of first UC-related complication until end of study (Week 96), whichever came first
  Time to UC-related complication starting when a participant reaches their assigned treatment target, compared between treatment target groups 1 and 2.
Difference in Time to UC-related Complication Compared Between Treatment Target Groups 2 and 3. | From date of treatment target achievement until date of first UC-related complication until end of study (Week 96), whichever came first
  Time to UC-related complication starting when a participant reaches their assigned treatment target, compared between treatment target groups 2 and 3.
Difference in time to UC-related complication compared between subgroups | From date of treatment target achievement until date of first UC-related complication until end of study (Week 96), whichever came first
  Time to UC-related complication compared between subgroups on and off corticosteroids at the time of achieving other relevant components of the treatment target.
Difference in Time to Achieve Treatment Target | up to 96 weeks
  Time taken to achieve the respective targets among the randomized groups. Time will be censored for subjects who do not achieve their assigned target by Week 48.
Fecal Calprotectin Levels | Baseline, weeks 8, 16, 32, 48, and 96.
  Change in fecal calprotectin levels from baseline to Weeks 8, 16, 32, 48, and 96.
C-Reactive Protein Concentration | Baseline, weeks 8, 16, 32, 48, 64, 80, and 96
  Change in C-Reactive Protein concentration from baseline to Weeks 8, 16, 32, 48, 64, 80, and 96.
Difference in time to UC-related complication (as in the primary outcome and secondary outcomes 2 and 3) | Up to week 96
  Time to UC-related complication (as in the primary outcome and secondary outcomes 2 and 3) in the subgroup of subjects who exclusively reach their assigned target and not a higher target by Week 48.
Evaluate the time to each type of UC-related complication | Up to week 96
  Evaluate, across the 3 target achievement groups, the time to each type of UC-related complication that comprises the primary endpoint.
Assess the effect of treatment(s) on UC-related complications | Up to week 96
  Assess the effect of treatment(s) on UC-related complications that is mediated through treatment targets.
Evaluate change in the UC-100 score from baseline to Weeks 16, 32, 48, and 96 | Up to week 96
  To evaluate change in the UC-100 score from baseline to Weeks 16, 32, 48, and 96 (both in the full and the achieved-target populations). The UC-100 is a composite disease activity index consisting of clinical, endoscopic, and histological findings.The total UC-100 score ranges from 1 to 100, with higher scores representing more severe disease activity.
Evaluate changes in the health-related quality of life (HRQoL) using the Inflammatory Bowel Disease Questionnaire (IBDQ) | Up to week 96
  To evaluate changes in the health-related quality of life (HRQoL) using the Inflammatory Bowel Disease Questionnaire (IBDQ) from baseline to all follow-up visits.The Inflammatory Bowel Disease Questionnaire (IBDQ) includes 32 questions on 4 domains of health-related quality of life (HRQoL); the total score ranges from 32 and 224, with a higher score signifying a better outcome.
Evaluate changes in the Work Productivity and Activity Impairment-UC (WPAI-UC) questionnaire | Up to week 96
  To evaluate changes in the Work Productivity and Activity Impairment-UC (WPAI-UC) questionnaire from baseline to all follow-up visits.The WPAI-UC (Work Productivity and Activity Impairment Questionnaire) consists of 6 questions that will grade the productivity while the participant is working on a scale from 0 to 10; a higher score signifies a higher impact on work productivity.
Evaluate the change in Mayo Clinic Score (MCS; and subcomponents including the MES) | Up to week 96
  To evaluate the change in Mayo Clinic Score (MCS; and subcomponents including the MES) from baseline to Week 16,32,48 and 96/end of study (EOS). The Mayo Clinic Score for Ulcerative Colitis is a score that ranges from 0 to 12 with higher scores indicating worse severity. The score has four items (Stool Frequency, Rectal Bleeding, Mucosal appearance at endoscopy, Physician rating of disease activity) each rated from 0 to 3, where 3 means highest severity.
Describe the change in Geboes scores from baseline to baseline to Week 16, 32, 48 and 96/end of study (EOS) | Up to week 96
  To describe the change in Geboes scores from baseline to baseline to Week 16, 32, 48 and 96/end of study (EOS). Geboes score is the most commonly used histological score in ulcerative colitis [UC] and is divided in 6 grades: architectural changes [grade 0], chronic inflammatory infiltrate [grade 1], lamina propria neutrophils and eosinophils [grade 2], neutrophils in epithelium [grade 3], crypt destruction [grade 4] and erosions or ulcerations [grade 5].
Describe the change in RHI scores from baseline to all baseline to Week 16, 32, 48 and 96/end of study (EOS) | Up to week 96
  To describe the change in RHI scores from baseline to all baseline to Week 16, 32, 48 and 96/end of study (EOS). The Robarts Histopathology Index (RHI) is a validated instrument that measures histological disease activity in ulcerative colitis. The RHI assesses four characteristics of mucosal activity, inflammatory infiltrate, lamina propria neutrophils, neutrophils in epithelium, and erosion or ulceration, all of which are rated on a scale of 0 to 3, with higher scores representing more severe disease activity.
Describe the change in Nancy Histological Index scores from baseline to baseline to Week 16, 32, 48 and 96/end of study (EOS) | Up to week 96
  To describe the change in Nancy Histological Index scores from baseline to baseline to Week 16, 32, 48 and 96/end of study (EOS). The Nancy Histological Index is made up of 3 items: acute inflammatory cell infiltrates, chronic inflammatory cell infiltrates, and the presence of ulceration. Histological disease activity is graded on a 5-point scale; from grade 0 (no histologically significant disease) to grade 4 (severely active disease), with this grade being determined by the scoring algorithm.
Evaluate the numbers of AEs and SAEs among the 3 randomized groups | Up to week 96
  To evaluate the numbers of AEs and SAEs among the 3 randomized groups.
Validate the Symptoms and Impacts Questionnaire for UC (SIQ-UC) tool in English-fluent subjects | Up to week 96
  To validate the Symptoms and Impacts Questionnaire for Ulcerative Colitis (SIQ-UC) tool in English-fluent subjects. SIQ-UC consists of a symptom domain, which includes Gastrointestinal, pain and discomfort, nutrition-related, and fatigue-related symptoms; and an impact domain, which includes concepts related to daily activities, nutrition, emotional well-being, and productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Jairath, MD, Principal Investigator — Alimentiv Inc.
Locations (58):
- United States (5):
  - St. Joseph Mercy Hospital/Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Icahn School of Medicine at Mt Sinai Hospital, New York, New York
  - New York-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Digestive Health Partners - Asheville Gastroenterology Associate, Asheville, North Carolina
  - Atrium Health (Carolinas HealthCare), Charlotte, North Carolina
- Belarus (2):
  - Gomel Regional Clinical Hospital, Homyel, Homiel
  - Vitebsk Regional Clinical Hospital, Vitebsk, Vitebsk Oblast
- Belgium (3):
  - Imelda Ziekenhuis Bonheiden, Bonheiden, Antwerp
  - University Hospital Ghent, Ghent, East Flanders
  - UZ Leuven - University Hospital Gasthuisberg, Leuven, Flemish Brabant
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - GIRI (GI Research Institute), Vancouver, British Columbia
  - Barrie GI Associates Inc., Barrie, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre - University Campus, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - ABP Research Services Corp., Oakville, Ontario
  - Taunton Surgical Centre, Oshawa, Ontario
  - Toronto Immune and Digestive Health Institute (TIDHI), Toronto, Ontario
  - McGill University Health Centre (MUHC) Montreal General Hospital, Montreal, Quebec
- France (6):
  - CH Saint Etienne Hopital Nord, Saint-Priest-en-Jarez, Auvergne-Rhône-Alpes
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Bourgogne-Franche-Comté
  - CHRU De Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy, Grand Est
  - CHRU de Lille - Hopital Claude Huriez, Lille, Hauts-de-France
  - CHU de Bordeaux - Hopital Haut Leveque - Groupe Hospitalier Sud, Pessac, Nouvelle-Aquitaine
  - CHRU Montpellier - Hopital Saint Eloi, Montpellier, Occitanie
- Italy (5):
  - Azienda Ospedaliera - Polyclinico Sant'Orsola-Malpighi, Bologna, Emilia-Romagna
  - Ospedale San Raffaele S.r.I., Milan, Milan
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Azienda Ospedaliera di Padova, Padua, Padua
  - Policlinico Universitario Agostino Gemelli, Roma, Rome
- Netherlands (4):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Catharina Hospital, Eindhoven, North Brabant
  - ETZ Hospital Tilburg, Tilburg, North Brabant
  - Amsterdam UMC - Academisch Medisch Centrum, Amsterdam, North Holland
- Poland (8):
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - GASTROMED - Kopon, Zmudzinski I Wspolnicy Sp.j., Torun, Kuyavian-Pomeranian Voivodeship
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow, Lesser Poland Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z.o.o., Sopot, Pomeranian Voivodeship
  - Sonomed Sp. z o.o. - Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Szpital Miejski Sw. Jana Pawla II w Elblagu, Elblag
  - Oddział Gastroenterologiczny SP ZOZ w Łęcznej, Łęczna
- Ukraine (7):
  - Dniepropetrovsk State Medical Academy, Dnipro
  - Odesa Regional Clinical Hospital, Odesa
  - Ternopil City Communal Emergency Medical Care Hosp, Ternopil
  - Uzhhorod National University, Uzhhorod
  - Vinnytsia City Clinical Hospital #1, Dept of Gastroenterology, Vinnytsia
  - Vinnytsia M.I. Pyrohov Regional Clinical Hospital, Vinnytsia
  - City Clinical Hospital #9 Dept of Gastrosurgery SI Zaporizhzhia MA of PGE of MoHU, Zaporizhzhia
- United Kingdom (8):
  - Hampshire Hospitals NHS Foundation Trust - The Royal Hampshire County Hospital, Winchester, Hampshire
  - Oxford University Hospitals NHS Foundation - John Radcliffe Hospital, Headington, Oxford
  - University Hospitals Birmingham NHS Foundation Trust (UHB) - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Russells Hall Hospital, Dudley, West Midlands
  - Hull & East Yorkshire NHS Trust, Hull, Yorkshire
  - Barts Health NHS Trust / Whipps Cross University Hospital, Leytonstone
  - Barts Health NHS Trust - Royal London Hospital, London
  - University of Nottingham NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jairath V, Zou G, Wang Z, Adsul S, Colombel JF, D'Haens GR, Freire M, Moran GW, Peyrin-Biroulet L, Sandborn WJ, Sebastian S, Travis S, Vermeire S, Radulescu G, Sigler J, Hanzel J, Ma C, Sedano R, McFarlane SC, Arya N, Beaton M, Bossuyt P, Danese S, Green D, Harlan W 3rd, Horynski M, Klopocka M, Petroniene R, Silverberg MS, Wolanski L, Feagan BG. Determining the optimal treatment target in patients with ulcerative colitis: rationale, design, protocol and interim analysis for the randomised controlled VERDICT trial. BMJ Open Gastroenterol. 2024 Feb 8;11(1):e001218. doi: 10.1136/bmjgast-2023-001218. PMID 38336367
- See also: Determining the optimal treatment target in patients with ulcerative colitis: rationale, design, protocol and interim analysis for the randomised controlled VERDICT trial — https://bmjopengastro.bmj.com/content/11/1/e001218